CLINICAL TRIAL: NCT05956262
Title: The Effect of Portable AR on Tooth Brushing Skill for Elementary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20200073
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Augmented reality; dental plaque; schoolchildren
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR group (Experimental): Student in AR group received a two-time repeated AR-based training for 30 minutes at two-week intervals.
  Interventions: Device: AR-toothbrush machine
- traditional group (Experimental): Students in the traditional group received a two-time repeated 10-minute lesson regarding proper toothbrushing skills in the classroom at two-week intervals.
  Interventions: Behavioral: Teach proper brushing skills

INTERVENTIONS:
Device: AR-toothbrush machine — Student in AR group received a two-time repeated AR-based training for 30 minutes at two-week intervals. The AR-based training system (PVIX Oral, EPED) digitized the steps of the toothbrushing technique applying optical tracking technology to enable the participants to obtain immediate scoring after the completion of practice. The scoring depends on the level of removing simulated dental plaque. The AR system was equipped with an optical tracking unit, a 3D training head model, and a wireless toothbrush. The toothbrushing practice time for the upper and lower jaw is 3 minutes, respectively. A tooth-brushing song played while the students implemented.
  Arms: AR group
Behavioral: Teach proper brushing skills — Students in the traditional group received a two-time repeated 10-minute lesson regarding proper toothbrushing skills in the classroom at two-week intervals. The students were taught by a well-trained dental hygienist using teaching aids (such as dental models, and toothbrushes).
  Arms: traditional group

SUMMARY:
The aim of this study An augmented reality (AR) simulation toothbrushing machine was developed to train proper brushing technique for children. The investigators aimed to evaluate the effects of AR brushing machine on knowledge of dental clearing skill, self-efficacy and dental plaque control in elementary schoolchildren in Taiwan.

DETAILED DESCRIPTION:
A quasi-experimental design was conducted; ten intervention schools (AR group) and ten comparison schools were selected from elementary schools. Overall, grade 3-6 students in the AR group (n = 290) and the traditional group (n = 311), respectively. Students in the AR group received a two-time repeated AR-based training for 30 minutes at two-week intervals. Students in the CG received traditional classroom-based teaching. Baseline and follow-ups information was collected using dental plaque examinations and questionnaires. The generalized estimating equations(GEE) were used to evaluate the outcomes between two groups over time.

ELIGIBILITY:
Inclusion Criteria:

* Primary school students 3 to 6 grades

Exclusion Criteria:

* Schoolchildren with disability certification.
* Schoolchildren with congenital severe oral diseases (eg. cleft lip and palate )
* Disability to operate the AR system

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 601 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) | Change from Baseline at 2-week after intervention
  Each tooth is divided into six surfaces, and the PCR record is calculated ( range 0-100% )
Plaque Control Record (PCR) | Change from Baseline at 4-week after intervention
  Each tooth is divided into six surfaces, and the PCR record is calculated ( range 0-100% )
Self-efficacy | Change from Baseline at 2-week after intervention
  2 questions , e.g: I feel confident.Response 1 = strongly disagree 2 = Disagree 3 = Normal 4 = agree 5 = strongly agree
Self-efficacy | Change from Baseline at 4-week after intervention
  2 questions , e.g: I feel confident.Response 1 = strongly disagree 2 = Disagree 3 = Normal 4 = agree 5 = strongly agree
Skill of Toothbrushing | Change from Baseline at 2-week after intervention
  5 questions , e.g: The toothbrush is pressed against the gums at a 45-degree angle.Response multiple choice
Skill of Toothbrushing | Change from Baseline at 4-week after intervention
  5 questions , e.g: The toothbrush is pressed against the gums at a 45-degree angle.Response multiple choice

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan